CLINICAL TRIAL: NCT00376064
Title: A Multicenter, Single Arm, Proof of Concept Study to Investigate the Efficacy of an 8 Month Combination Therapy of Octreotide and Cabergoline in Acromegalic Patients Only Partially Responsive to Somatostatin Analog Monotherapy
Brief Title: Efficacy of Octreotide Acetate and Cabergoline in Patients With Acromegaly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSMS995BDE16
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2011-09

CONDITIONS: Acromegaly
Keywords: Growth hormone (GH); IGF-1; Acromegaly; Pituitary adenoma; Brain tumor; Brain cancer; Octreotide acetate
MeSH Terms: conditions — Acromegaly; Pituitary Neoplasms; Brain Neoplasms | interventions — Octreotide; Cabergoline; pegvisomant

ARMS (1):
- SMS995 + Carbegolin, Somavert + SMS995 (Experimental)
  Interventions: Drug: Octreotide acetate and cabergoline/Octrotide and Somavert

INTERVENTIONS:
Drug: Octreotide acetate and cabergoline/Octrotide and Somavert

SUMMARY:
This study will investigate the efficacy of a combination treatment with octreotide acetate and cabergoline in acromegalic patients that are only partially responsive to a somatostatin analog monotherapy

ELIGIBILITY:
Inclusion criteria:

* Male and female patients (> 18 years) with prior surgery of micro- or macroadenoma of the pituitary.
* At least 6 months chronic treatment with 30mg octreotide (long acting release).
* Partial responsiveness, which is defined as follows: at any one point within the 6 months monotherapy with 30mg/month octreotide (long acting release) the patient must have experienced a decrease in GH and IGF-1 of at least 25% as compared to pre-monotherapy values (= baseline). Note: For efficacy analysis GH- and IGF-1-values measured in the central laboratory at visit 1 (=study baseline) will be used.
* Lack of suppression of GH nadir to < 1.0 µg/L, after oral administration of 75 g of glucose (OGTT) and IGF-I levels at least 10% above the normal value ± 2 SD (adjusted for age and gender; Brabant 2003) must be proven within 4 weeks prior to visit 1. However, if acromegaly symptoms are inadequately controlled as defined in the acromegaly comorbidities and symptom evaluation (as judged by the investigator), an abnormal GH or IGF-1-value as defined above is sufficient.
* Patient's written informed consent.

Exclusion criteria:

* Requires surgery for recent significant deterioration in visual fields or other neurological signs, which are related to the pituitary tumor mass.
* Radiotherapy planned or radiotherapy for acromegaly within the last 2 years.
* Symptomatic cholelithiasis that is clinically relevant.
* Receiving treatment with dopamine agonists within the last 6 months or prior treatment with GH-receptor-antagonists.
* Patients with renal insufficiency, Raynaud-Syndrome or gastrointestinal ulcer/ bleeding cannot be included in the study or psychose in anamnesis.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-03; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Biochemical control (% of patients) as measured by GH- and IGF-1-values (baseline, EOS) | 8 months

SECONDARY OUTCOMES:
Effect of tumor size | 8 months
Biochemical control (mean, normalization) as measured by GH- and/or IGF-1-values | 8 months
Control clinical of symptoms of acromegaly | 8 months
Quality of Life assessment | 8 months
Safety and tolerability as assessed by frequency of AEs | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (16):
- Germany (16):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Würzburg